CLINICAL TRIAL: NCT01881854
Title: Cross Sectional Study of Sleep-wake and Melatonin Patterns in Patients Treated for Craniopharyngiomas Compared to Matched Controls
Brief Title: Sleep Wake and Melatonin Pattern in Craniopharyngioma
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, chief physician, Rigshospitalet, Denmark
Other Study IDs: Cranio-sleep-melatonin
Record Dates: First submitted 2013-06-12; First posted 2013-06-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Sleep Disorders, Circadian Rhythm; Craniopharyngioma
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Craniopharyngioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- craniopharyngioma: Patients treated for craniopharyngioma, most of them on pituitary substitution therapy
- Healthy controls: matched for gender, age and BMI to the patients

SUMMARY:
The hypothalamus is a part of the brain containing a number of nuclei with a variety of functions. It is central in the regulation of hormone secretion, sleep, and circadian functions. The suprachiasmatic nucleus of the hypothalamus is a key component in controlling circadian rhythms and generates the rhythm of melatonin secretion from the pineal gland and cortisol secretion. Both melatonin and cortisol are involved in the regulation of circadian rhythms and sleep.

Craniopharyngiomas are a type of brain tumors that usually affect the hypothalamus indirectly. In general, they are locally aggressive invading crucial structures e.g. the hypothalamus, the pituitary, and the optic nerve. Compared to healthy controls, craniopharyngioma patients have previously been reported with impaired quality of life, increased self-reported general and physical fatigue, increased daytime sleepiness, and increased prevalence of severe sleepiness

Damage to the hypothalamus by local tumour or its treatment might involve the suprachiasmatic nucleus and thereby melatonin secretion leading to disturbed circadian function causing clinical manifestations in terms of daytime sleepiness and fatigue.

The investigators aimed to assess the influence of craniopharyngiomas or their treatment on melatonin secretion, and the association with sleep pattern, sleep quality, fatigue, and sleepiness.

15 patients with craniopharyngioma and 15 gender, age, and BMI matched healthy controls were included. Salivary melatonin and cortisol were measured over a 24h-period. Sleep-wake patterns were characterized by two weeks of actigraphy recordings and sleep diaries. Sleepiness, fatigue, sleep quality, and general health were assessed by questionnaires.

DETAILED DESCRIPTION:
The hypothalamus is a part of the brain containing a number of nuclei with a variety of functions. It is central in the regulation of hormone secretion, sleep, and circadian functions. The suprachiasmatic nucleus of the hypothalamus is a key component in controlling circadian rhythms and generates the rhythm of melatonin secretion from the pineal gland and cortisol secretion. Both melatonin and cortisol are involved in the regulation of circadian rhythms and sleep.

Craniopharyngiomas are a type of brain tumors that usually affect the hypothalamus indirectly. In general, they are locally aggressive invading crucial structures e.g. the hypothalamus, the pituitary, and the optic nerve. Compared to healthy controls, craniopharyngioma patients have previously been reported with impaired quality of life, increased self-reported general and physical fatigue, increased daytime sleepiness, and increased prevalence of severe sleepiness

Damage to the hypothalamus by local tumour or its treatment might involve the suprachiasmatic nucleus and thereby melatonin secretion leading to disturbed circadian function causing clinical manifestations in terms of daytime sleepiness and fatigue.

The investigators aimed to assess the influence of craniopharyngiomas or their treatment on melatonin secretion, and the association with sleep pattern, sleep quality, fatigue, and sleepiness.

15 patients with craniopharyngioma and 15 gender, age, and BMI matched healthy controls were included. Salivary melatonin and cortisol were measured over a 24h-period. Sleep-wake patterns were characterized by two weeks of actigraphy recordings and sleep diaries. Sleepiness, fatigue, sleep quality, and general health were assessed by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients treated for former craniopharyngiomas
* aged 18-70 years.

Exclusion Criteria:

* insufficient substitution of pituitary hormone deficiencies within six months prior to inclusion
* total blindness
* clinically significant liver or renal disease
* use of non-steroid anti-inflammatory drugs
* beta-receptor antagonists
* antidepressants that affect serotonin
* active cancer
* epileptic seizures
* working night-shift
* breast feeding
* pregnancy,
* alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated for craniopharyngioma with surgery and some also irradiation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
24h melatonin and cortisol concentrations | 1 year

SECONDARY OUTCOMES:
actigraphy | 1 year
  Measuring daily activity by actigraph measurements

OTHER OUTCOMES:
sleep-wake characteristics | 1 year
  Sleep-wake pattern of individual participants measured by diaries

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: Undecided